CLINICAL TRIAL: NCT00054639
Title: A Phase II Study of G3139 (Bcl-2 Antisense) And Rituximab in Patients With Recurrent B-cell Non-Hodgkinâs Lymphomas
Brief Title: Oblimersen Sodium and Rituximab in Treating Patients With Recurrent B-cell Non-Hodgkin Lymphoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2011-00617; ID02-148; N01CM17003 (NIH); N01CM62202 (NIH); N01CM17107 (NIH); N01CM62203 (NIH); NCT01654952 (obsolete NCT alias)
Record Dates: First submitted 2003-02-05; First posted 2003-02-06 (Estimated); Results first posted 2011-02-21 (Estimated); Last update posted 2014-05-28 (Estimated); Status verified 2013-03

CONDITIONS: Cutaneous B-cell Non-Hodgkin Lymphoma; Extranodal Marginal Zone B-cell Lymphoma of Mucosa-associated Lymphoid Tissue; Intraocular Lymphoma; Nodal Marginal Zone B-cell Lymphoma; Recurrent Adult Burkitt Lymphoma; Recurrent Adult Diffuse Large Cell Lymphoma; Recurrent Adult Diffuse Mixed Cell Lymphoma; Recurrent Adult Diffuse Small Cleaved Cell Lymphoma; Recurrent Adult Grade III Lymphomatoid Granulomatosis; Recurrent Adult Immunoblastic Large Cell Lymphoma; Recurrent Adult Lymphoblastic Lymphoma; Recurrent Grade 1 Follicular Lymphoma; Recurrent Grade 2 Follicular Lymphoma; Recurrent Grade 3 Follicular Lymphoma; Recurrent Mantle Cell Lymphoma; Recurrent Marginal Zone Lymphoma; Recurrent Small Lymphocytic Lymphoma; Small Intestine Lymphoma; Splenic Marginal Zone Lymphoma; Testicular Lymphoma; Waldenström Macroglobulinemia
MeSH Terms: conditions — Intraocular Lymphoma; Lymphoma, B-Cell, Marginal Zone; Burkitt Lymphoma; Lymphoma, Large B-Cell, Diffuse; Lymphoma, Non-Hodgkin; Lymphoma, Large-Cell, Immunoblastic; Precursor Cell Lymphoblastic Leukemia-Lymphoma; Lymphoma, Follicular; Lymphoma, Mantle-Cell; Leukemia, Lymphocytic, Chronic, B-Cell; Waldenstrom Macroglobulinemia | interventions — oblimersen; Rituximab

ARMS (1):
- Treatment (oblimersen sodium and monoclonal antibody therapy) (Experimental): Patients receive oblimersen sodium IV continuously on days 1-7, 15-21, and 29-35 and rituximab IV over 4-6 hours on days 3, 8, 15, 22, 29, and 36. Patients achieving stable disease or objective response may receive one additional course of treatment.
  Interventions: Biological: oblimersen sodium; Biological: rituximab; Other: laboratory biomarker analysis

INTERVENTIONS:
Biological: oblimersen sodium — Given IV
  Other Names: augmerosen; G3139; G3139 bcl-2 antisense oligodeoxynucleotide; Genasense
Biological: rituximab — Given IV
  Other Names: IDEC-C2B8; IDEC-C2B8 monoclonal antibody; Mabthera; MOAB IDEC-C2B8; Rituxan
Other: laboratory biomarker analysis — Correlative studies

SUMMARY:
The goal of this clinical research study is to learn if the combination of oblimersen sodium and rituximab can help to shrink or slow the growth of the tumor in patients with B-cell non-Hodgkin's lymphoma who have not responded to earlier treatment. Oblimersen Sodium is an investigational drug. The safety of this combination treatment will also be studied

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine the therapeutic efficacy and toxicity of G3139 (oblimersen sodium) and Rituximab in patients with recurrent B-cell NHL.

SECONDARY OBJECTIVES:

I. To determine the effect of G3139 and Rituximab on the level of Bcl-2 expression.

II. The secondary objective of this study is to evaluate the effect of G3139 and Rituximab on Bcl-2 protein gene expression.

OUTLINE:

Patients receive oblimersen sodium intravenously (IV) continuously on days 1-7, 15-21, and 29-35 and rituximab IV over 4-6 hours on days 3, 8, 15, 22, 29, and 36. Patients achieving stable disease or objective response may receive one additional course of treatment.

After completion of study treatment, patients are followed up every 3 months.

ELIGIBILITY:
Inclusion Criteria:

* Must have recurrent B-cell NHL and measurable disease
* No anti-lymphoma therapy within the past 4 weeks
* Must have a good performance status (less than or equal to 2 Zubrod, greater than or equal to 60 Karnofsky)
* Absolute neutrophil count (ANC) greater than or equal to 1,000
* Platelets greater than or equal to 75,000
* Hemoglobin greater than or equal to 10 g/dL
* Bilirubin less than or equal to 1.5 mg/dL
* Serum glutamic oxaloacetic transaminase (SGOT), serum glutamic pyruvate transaminase (SGPT) less than or equal to 2 times upper limit of laboratory normals
* Alkaline phosphatase less than or equal to 2 times upper limit of laboratory normals
* Serum creatinine less than or equal to 1.8 mg/dL
* Must sign a consent form, and must have a life expectancy of greater than 12 weeks
* No more than 3 prior chemotherapy regimens
* Patients who are either Rituximab naive, have previously responded to Rituximab, or are refractory to Rituximab used alone or in combination with chemotherapy

Exclusion Criteria:

* Human immunodeficiency virus (HIV) positive
* Active infection or history of opportunistic infections
* Pregnant women and women of childbearing age who are not practicing adequate contraception; men who are not willing to use an effective method of contraception
* History of second cancer (except for adequately treated basal cell or squamous cell skin cancer, in situ cervical cancer or other cancer for which the patient has been disease-free for 5 or more years)
* Active autoimmune disease
* Other significant medical diseases
* Patients with chronic lymphocytic leukemia (CLL)
* Prior exposure to G3139

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2003-01; Primary Completion 2010-01 (Actual); Study Completion 2010-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Barbara Pro, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- M D Anderson Cancer Center, Houston, Texas, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment Period: January 07, 2003 to October 01, 2005. Recruitment was done at UT MD Anderson Cancer Center Clinics.
Pre-assignment Details: Two participants enrolled but not assigned were not included in baseline measures. Of the total 48 participants enrolled, 42 were evaluable for response and 46 for toxicity.
Groups:
- Oblimersen + Rituximab: Oblimersen 3 mg/kg/day continuous intravenous infusion daily for 7 days on alternated weeks on week 1, 3 and 5 (days 1 through 7, 15 through 21, and 29 through 35); Rituximab 375 mg/m2 intravenous infusion for six doses on days 3, 8,15, 22, 29, and 36.
Period: Overall Study
Arm/Group | Oblimersen + Rituximab
Started | 48
Completed | 46
Not Completed | 2
Not completed — Lack of Efficacy | 1
Not completed — Physician Decision | 1

BASELINE CHARACTERISTICS:
Arm/Group | Oblimersen + Rituximab
Number analyzed (Participants) | 46
Age, Continuous [Median (Full Range); unit: years] | 59 [35 to 82]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 33
  Male | 13
Region of Enrollment [Number; unit: participants]
  United States | 46

OUTCOME MEASURES:

1. Primary Outcome: Number of Patients With Objective Response
Description: Efficacy as measured by objective response complete (CR) and partial (PR) response rates at 2 months following study treatment
Time Frame: 2 months following study treatment
Population: Analysis was per protocol. Of the 48 participants enrolled, only 42 were evaluable for response.
Measure: Number; unit: participants
Arm/Group | Oblimersen + Rituximab
Number analyzed (Participants) | 42
participants
  Complete Responses | 10
  Partial Responses | 8

ADVERSE EVENTS:
Time Frame: 2 Years, 10 Months
Arm/Group | Oblimersen + Rituximab
Serious Adverse Events (participants affected / at risk) | 15/46
Other Adverse Events (participants affected / at risk) | 46/46
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Oblimersen + Rituximab (N=46)
Anaemia (Blood and lymphatic system disorders) | 1 (1)
Thrombocytopenia (Blood and lymphatic system disorders) | 2 (2)
Neutropenia (Blood and lymphatic system disorders) | 7 (7)
Fatigue (General disorders) | 3 (3)
Oedema (Eye disorders) | 1 (1)
Fever (Infections and infestations) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Oblimersen + Rituximab (N=46)
Anaemia (Blood and lymphatic system disorders) | 23 (23) — Grade 1 and 2
Thrompbocytopenia (Blood and lymphatic system disorders) | 8 (8) — Grades 1 and 2
Neutropenia (Blood and lymphatic system disorders) | 3 (3) — Grades 1 and 2
Fatigue (Gastrointestinal disorders) | 17 (17) — Grades 1 and 2
Odema (Eye disorders) | 9 (9) — Grades 1 and 2
Rash (Skin and subcutaneous tissue disorders) | 9 (9) — Grades 1 and 2
Fever (Infections and infestations) | 5 (5) — Grades 1 and 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less